CLINICAL TRIAL: NCT06324058
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study Evaluating the Safety and Efficacy of Cryoablation Versus BCG Instillation Therapy for High-risk NMIBC
Brief Title: Cryoablation Versus BCG Instillation Therapy for High-risk NMIBC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Haowen Jiang, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huashan_H
Record Dates: First submitted 2024-03-10; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Transurethral Resection of Bladder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation group (Experimental): Transurethral resection of bladder tumor, instant cryoablation of the bladder tumor resection site.
  Interventions: Procedure: Transurethral cryoablation; Procedure: Transurethral resection of bladder tumor; Drug: Bcg Intravesical
- Control group (Active Comparator): Transurethral resection of bladder tumor, conventional BCG instillation after surgery
  Interventions: Procedure: Transurethral resection of bladder tumor; Drug: Bcg Intravesical

INTERVENTIONS:
Procedure: Transurethral cryoablation — Using an intracavitary cryoablation balloon, cryoablation is performed on the wound surface after tumor resection. The wound surface is frozen for 2 rounds, with each round lasting 3 minutes, to fully cover the wound surface.
  Arms: Cryoablation group
Procedure: Transurethral resection of bladder tumor — Resection of bladder tumor using resectoscopy, which is a standard procedure to treat non-muscle invasive bladder cancer
  Other Names: TURBt
Drug: Bcg Intravesical — Bacillus Calmette-Guerin instillation of bladder after surgery according to the NCCN bladder cancer guidelines. At least 6 weeks induction instillation is required for high-risk NMIBC patients. At least 1 year maintenance instillation is recommended.

SUMMARY:
This trial plans to enroll 190 eligible patients and randomize them into two groups with a 1:1 ratio, with 95 patients in each group. The experimental group will receive immediate cryoablation therapy at the resection site after TUR, while the control group will only undergo TUR and receive conventional BCG instillation therapy postoperatively. Both groups of subjects will undergo Re-TURBT or cystoscopy 10-12 weeks after surgery to compare the tumor-free residual rates and adverse events between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 85, male or female;
2. Preoperatively diagnosed with T1 stage or meeting the criteria for high-risk bladder cancer (accord with the "2023 NCCN Bladder Cancer Guidelines");
3. Good compliance and able to cooperate with observation;
4. Able to understand the purpose of the trial, agree to participate in this study, and have signed the informed consent form.

Exclusion Criteria:

1. Patients with severe infectious diseases such as bacteremia and toxemia;
2. Patients with severe coagulation dysfunction;
3. Patients with severe heart, brain, lung, liver, kidney and other diseases who cannot tolerate surgery;
4. Patients with other concurrent malignancies;
5. Postoperative pathological diagnosis of bladder cancer patients in Tis, Ta, or T2 stages;
6. Preoperative CT/MRI assessment showing tumor invasion beyond the bladder (T3 stage or above);
7. Preoperative assessment indicating distant metastasis or enlarged pelvic lymph nodes;
8. Pregnant or breastfeeding women;
9. Other situations assessed by researchers as unsuitable for inclusion in this study, such as inappropriate anatomical structure, mental or psychological disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-03-18 (Estimated); Primary Completion 2025-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Tumor residual rate | 10-12 weeks after initial TURBt
  10-12 weeks after the initial TUR, Re-TUR or cystoscopy is performed on the original resection site, and a biopsy of the tissue at the original resection site is conducted to analyze and observe whether there is any tumor residue at the original tumor site.

SECONDARY OUTCOMES:
Recurrence | 2 years
  Non-muscle invasive bladder cancer recurrence during follow-up
Progression | 2 years
  Muscle invasive bladder cancer recurrence during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Haowen Jiang, Pro., Principal Investigator — Huashan Hospital

IPD SHARING:
Plan to Share IPD: No